CLINICAL TRIAL: NCT01491503
Title: Open Label, Randomized, 6-sequence Crossover Study to Evaluate the Drug-drug Interaction Between Montelukast Sodium and Levocetirizine Dihydrochloride in Health Male Volunteers
Brief Title: A Drug Interaction Study of Montelukast and Levocetirizine
Acronym: MOLZ
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-MOLZ-101
Record Dates: First submitted 2011-10-14; First posted 2011-12-14 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Healthy
Keywords: montelukast; levocetirizine; interaction
MeSH Terms: interventions — levocetirizine; montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Montelukast and levocetirizine (Experimental)
  Interventions: Drug: Montelukast & levocetirizine
- Montelukast (Active Comparator)
  Interventions: Drug: montelukast sodium
- Levocetirizine (Active Comparator)
  Interventions: Drug: Levocetirizine

INTERVENTIONS:
Drug: Levocetirizine — Levocetirizine dihydrochloride 5mg. PO. Single dose.
  Arms: Levocetirizine
Drug: montelukast sodium — Montelukast sodium 10mg. PO. Single dose.
  Arms: Montelukast
Drug: Montelukast & levocetirizine — Montelukast sodium 10mg & levocetirizine dihydrochloride 5mg PO. Single dose.
  Arms: Montelukast and levocetirizine

SUMMARY:
The purpose of this study is to evaluate the drug-drug interaction between montelukast sodium and levocetirizine dihydrochloride in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male
* Age between 20 and 55
* Signed informed consent

Exclusion Criteria:

* Has a history of hypersensitivity to IP ingredients
* Hypotension or hypertension
* Has a history of acute infection within 14days of screening

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
AUClast | 0-36hrs
Cmax | 0-36hrs

SECONDARY OUTCOMES:
Tmax | 0-36hrs
T1/2 | 0-36hrs
AUCinf | 0-36hrs

CONTACTS AND LOCATIONS:
Overall Officials: Wooseong Huh, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung medical center, Seoul, South Korea